CLINICAL TRIAL: NCT04380558
Title: Prevalence and Consequences of Urinary Incontinence in People with Chronic Pulmonary Diseases Referred for Pulmonary Rehabilitation
Acronym: PRECUI-PR
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: PRECUI-PR
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pulmonary Disease; Pulmonary Rehabilitation; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective observational cohort: Every patient referred to pulmonary rehabilitation program will be eligible. They will will be asked to answer two questionnaires about urinary incontinence symptoms (see outcomes) to assess the prevalence and the type of these symptoms.
  They will subsequently participate in their usual pulmonary rehabilitation program consisting in 90min sessions (including endurance training, muscle strengthening and self-management), 3x/week for 8weeks (centre 1) or 2x60min sessions (including the same components), 3x/week for 8weeks (centre 2).
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Patients will be asked to answer two questionnaires about urinary incontinence symptoms (see outcomes) to assess the prevalence and the type of these symptoms.
  They will subsequently participate in their usual pulmonary rehabilitation program consisting in 90min sessions (including endurance training, muscle strengthening and self-management), 3x/week for 8weeks (centre 1) or 2x60min sessions (including the same components), 3x/week for 8weeks (centre 2).

SUMMARY:
Urinary incontinence is a frequent chronic condition in general population. It is even more frequent in people with chronic respiratory disease due to several factors, including but not limited to frequent cough. Urinary incontinence may be more frequent during exercise so that it may contribute to the general deconditioning associated with chronic respiratory disease.

Although pulmonary rehabilitation is a cornerstone in the management of people with chronic respiratory disease to break this spiral of worsening dyspnea, little is known about the prevalence of urinary incontinence among those people referred for pulmonary rehabilitation nor about its impact on the effects of the program.

DETAILED DESCRIPTION:
Experimental design:

People referred for pulmonary rehabilitation in two centres will be offer to participate in the study. Those people who will agree to participate and give their formal consent will be asked to answer two questionnaires about urinary incontinence symptoms (see outcomes) to assess the prevalence and the type of these symptoms.

They will subsequently participate in their usual pulmonary rehabilitation program consisting in 90min sessions (including endurance training, muscle strengthening and self-management), 3x/week for 8weeks (centre 1) or 2x60min sessions (including the same components), 3x/week for 8weeks (centre 2).

The effects of the pulmonary rehabilitation program on usual clinical outcomes (according to each centre routine practice; tests may differ between centres) will be compared between those people with or without urinary incontinence symptoms.

As no prevalence data about urinary incontience was available at the time of study design, we planned to recruit the first 100 participants within the first year and to update the sample size calculation based on these preliminary data.

Among the 70 people actually included, 21 (30%) experienced urinary incontinence. Therefore, assuming a true prevalence of 30% in this population and a total width for the 95% confidence interval of 10%, we planned to recruit a total 341 participants.

The ethical approval to recruit this updated number of participants and to increase the duration of recruitment accordingly was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ans ;
* Referred for pulmonary rehabilitation ;

Non inclusion Criteria:

* History of pathology or prostate surgery ;
* Contra indication to pulmonary rehabilitation ;

Exclusion Criteria:

* Pregnant woman or likely to be ;
* Patient under guardianship ;
* Patient withdrawal ;
* Did not complete at least 18 pulmonary rehabilitation sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People reffered for pulmonary rehabilitation.
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of urinary incontinence symptoms | The questionnaire will be administered at baseline
  The prevalence of urinary incontinence symptoms will be assessed using the International Consultation on Incontinence Short Form
Prevalence of urinary incontinence symptoms | The questionnaire will be administered at the end of the program (8weeks)
  The prevalence of urinary incontinence symptoms will be assessed using the International Consultation on Incontinence Short Form

SECONDARY OUTCOMES:
Type of urinary incontinence symptoms | The questionnaire will be administered at baseline
  The type of urinary incontinence symptoms will be assessed using the Urinary Symptom Profile questionnaire.
Type of urinary incontinence symptoms | The questionnaire will be administered at the end of the program (8weeks)
  The type of urinary incontinence symptoms will be assessed using the Urinary Symptom Profile questionnaire.
Exercise capacity - Six-minute walk test (meters) | The test will be administered at baseline
  The six-minute walk test will be performed before and after the completion of the pulmonary rehabilitation program. In addition, the proportion of people who improve for more than 25meters will be compared between those people with or without urinary incontinence symptoms.
Exercise capacity - Six-minute walk test (meters) | The test will be administered at the end of the program (8weeks)
  The six-minute walk test will be performed before and after the completion of the pulmonary rehabilitation program. In addition, the proportion of people who improve for more than 25meters will be compared between those people with or without urinary incontinence symptoms.
Exercise capacity - Six-minute stepper test (steps) | The test will be administered at baseline
  The six-minute stepper test will be performed before and after the completion of the pulmonary rehabilitation program. In addition, the proportion of people who improve for more than 20steps will be compared between those people with or without urinary incontinence symptoms.
Exercise capacity - Six-minute stepper test (steps) | The test will be administered at the end of the program (8weeks)
  The six-minute stepper test will be performed before and after the completion of the pulmonary rehabilitation program. In addition, the proportion of people who improve for more than 20steps will be compared between those people with or without urinary incontinence symptoms.
Exercise capacity - Constant workload exercise testing | The test will be administered at baseline
  The constant workload exercise testing will be performed before and after the completion of the pulmonary rehabilitation program. In addition, the proportion of people who improve for more than 101sec will be compared between those people with or without urinary incontinence symptoms.
Exercise capacity - Constant workload exercise testing | The test will be administered at the end of the program (8weeks)
  The constant workload exercise testing will be performed before and after the completion of the pulmonary rehabilitation program. In addition, the proportion of people who improve for more than 101sec will be compared between those people with or without urinary incontinence symptoms.
Quality of life - Saint Georges Respiratory Questionnaire (ranging from 0 to 100, higher score indicates worst quality of life) | The questionnaire will be administered at baseline
  The questionnaire will be administered before and after the completion of the pulmonary rehabilitation program. In addition, the proportion of people who improve for more than 4points will be compared between those people with or without urinary incontinence symptoms.
Quality of life - Saint Georges Respiratory Questionnaire (ranging from 0 to 100, higher score indicates worst quality of life) | The questionnaire will be administered at the end of the program (8weeks)
  The questionnaire will be administered before and after the completion of the pulmonary rehabilitation program. In addition, the proportion of people who improve for more than 4points will be compared between those people with or without urinary incontinence symptoms.
Mood status - Anxiety | The questionnaire will be administered at baseline
  Anxiety will be assessed using the Hospital Anxiety and Depression Scale (ranging for 0 to 15, higher score indicates worst anxiety)
Mood status - Anxiety | The questionnaire will be administered at the end of the program (8weeks)
  Anxiety will be assessed using the Hospital Anxiety and Depression Scale (ranging for 0 to 15, higher score indicates worst anxiety)
Mood status - Depression | The questionnaire will be administered at baseline
  Depression will be assessed using the Hospital Anxiety and Depression Scale (ranging for 0 to 15, higher score indicates worst anxiety)
Mood status - Depression | The questionnaire will be administered at the end of the program (8weeks)
  Depression will be assessed using the Hospital Anxiety and Depression Scale (ranging for 0 to 15, higher score indicates worst anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: David Debeaumont, MD, Principal Investigator — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Antoine Cuvelier, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France.; Tristan Bonnevie, MsC, Study Chair — ADIR Association, Bois-Guillaume, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Francis-Edouard Gravier, PT, Study Chair — ADIR Association, Bois-Guillaume, France; Jean-François Muir, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; ADIR Association, Bois-Guillaume, France; Bouchra Lamia, Prof, PhD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Jean Quieffin, MD, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Guillaume Prieur, PT, MsC, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Clément Médrinal, PT, MsC, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France. Service de réanimation, Groupe Hospitalier du Havre, France
Locations (2):
- France (2):
  - ADIR Association, Bois-Guillaume
  - Groupe Hospitalier du Havre, Le Havre

IPD SHARING:
Plan to Share IPD: No